CLINICAL TRIAL: NCT00708773
Title: A Phase I Genotype-Directed Dose-Escalation Study of Irinotecan (NSC616348, CPT-11, Camptosar) in Patients With Advanced Solid Tumors
Brief Title: Genotype-Directed Dose-Escalation Study of Irinotecan in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13934B
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — 90 minute IV infusion once every 3 weeks.
  Dose will be based on sex and genotype determination.
  Other Names: CPT-11; Camptosar

SUMMARY:
Describe the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of irinotecan in cancer patients with advanced solid tumors with UGT1A1 6/6 and 6/7 genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor or lymphoma that is appropriate for treatment with irinotecan.
* 18 years or older
* ECOG performance status 0-1
* Life expectancy of greater than 12 weeks.
* Normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/μl
  * absolute neutrophil count ≥ 1,500/μl
  * platelets ≥ 100,000/μl
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional ULN (≤5 X ULN in patients with hepatic metastases)
  * creatinine within normal institutional limits OR
  * glomerular filtration rate ≥50 ml/min/1.73 m2 for patients with creatinine levels above institutional normal as calculated by the modified MDRD equation recommended by the National Kidney Disease Education Program
* Measurable or assessable disease.
* Able to understand and the willing to sign a written informed consent document.
* Women of child-bearing potential and men and their partners must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
* Patients with UGT1A1 genotype 6/6, 6/7, and 7/7. Patients with either one or two of the rare alleles (i.e., 5 allele and 8 allele), and carriers of the *6 allele will not be enrolled in the study. Patients will have blood drawn for genotyping upon signing the informed consent form for this study.
* Patients taking any statin therapy should interrupt the dosing of the statin for the 3 days before and after the administration of irinotecan at each cycle

Exclusion Criteria:

* Biologic therapy, chemotherapy, radiotherapy, or investigational agent within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Cannot be receiving any other investigational agents.
* Use of colony growth factor within 3 week prior to study entry.
* Post-transplant patients, as they may be subject to severe neutropenia.
* Uncontrolled brain metastases. Patients with brain metastases must have stable neurologic status off of steroids and anticonvulsants for at least 4 weeks and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because irinotecan is an agent with the potential for teratogenic or abortifacient effects. Breastfeeding should be stopped.
* HIV-positive patients, as patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* History of inflammatory bowel disease requiring therapy or patients with chronic diarrhea syndromes or paralytic ileus.
* Patients who have undergone a major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to start of therapy cannot participate.
* Patients with prior pelvic irradiation cannot participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 3 weeks
dose-limiting toxicity | 3 weeks

SECONDARY OUTCOMES:
pharmacokinetics | 3 weeks
anti-tumor response | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Federico Innocenti, MD, PhD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois